CLINICAL TRIAL: NCT00946569
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group Exploratory Study of the Safety and Efficacy of JNJ-39758979 in the Treatment of Adults With Persistent Asthma
Brief Title: A Study of the Safety and Effectiveness of JNJ-39758979 in the Treatment of Adults With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016423; 39758979ASH2001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: Asthma; Persistent asthma; Adults with persistent asthma; Chronic asthma; JNJ-39758979; Placebo
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment A (JNJ39758979) (Experimental): Participants will receive JNJ39758979 300mg once daily for 12 weeks.
  Interventions: Drug: JNJ39758979
- Treatment B (Placebo) (Placebo Comparator): Participants will receive matching placebo once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ39758979 — Participants will receive capsule-shaped tablet of JNJ39758979 300mg once daily orally for 12 weeks.
  Arms: Treatment A (JNJ39758979)
Drug: Placebo — Participants will receive matching placebo once daily orally for 12 weeks.
  Arms: Treatment B (Placebo)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of once daily oral administration of JNJ-39758979 in the treatment of adults (18 to 65 years of age) with persistent asthma.

DETAILED DESCRIPTION:
This is a multicenter, double-blind (neither physician nor participants knows the treatment that the participant receives), randomized (study medication is assigned by chance), placebo-controlled (an inactive substance is compared with a medication to test whether the medication has a real effect in a clinical study), parallel group (each group of participants will be treated at the same time), exploratory study (JNJ-39758979 is introduced in participants with asthma for the first time). This study consists of 4 phases: screening phase (4 weeks prior to the start of the run-in period), placebo run-in phase (2 weeks prior to the start of treatment phase), double-blind treatment phase (12 weeks), and posttreatment phase (5 weeks). Approximately 100 participants will be randomly allocated to 1 of 2 treatment groups: Treatment A (participants will receive JNJ-39758979 once daily) and treatment B (participants will receive placebo once daily). Safety will be evaluated by assessment of adverse events, clinical laboratory tests, vital signs, physical examination, and 12-lead electrocardiogram. Total study duration for each participant will be approximately 23 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of asthma for at least 6 months
* Short-acting beta-agonist use greater than or equal to 5 times in the 2 weeks prior to screening
* Healthy on the basis of physical examination, medical history, vital signs, and 12 lead ECG performed at screening
* Having adequate laboratory values
* No history of/active or latent tuberculosis
* Agree to use protocol defined contraceptive methods

Exclusion Criteria:

* History of life-threatening asthma attack requiring hospitalization for asthma within 5 years of screening, or emergency department treatment of asthma within the last month
* Moderate or severe renal insufficiency
* Cigarette smoking within the last year - Viral or bacterial vaccination within the last month (eg, FluMist)
* Human Immunodeficiency Virus (HIV) or Hepatitis B or C positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to Week 12 in pre-bronchodilator percent predicted Forced Expiratory Volume in 1 second (FEV1) value | Baseline (Week 0) and Week 12
  FEV1 will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. Lung volumes will be measured according to the body temperature, pressure, and saturated standard convention using the spirometer. Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol.

SECONDARY OUTCOMES:
Percent change from baseline in pre-bronchodilator percent predicted Forced Expiratory Volume in 1 second (FEV1) value | Week 1, Week 2, Week 4, and Week 8
  FEV1 will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. Lung volumes will be measured according to the body temperature, pressure, and saturated standard convention using the spirometer. Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol.
Percent change from baseline in post-bronchodilator percent predicted Forced Expiratory Volume in 1 second (FEV1) value | Week 4 and Week 12
  FEV1 will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. Lung volumes will be measured according to the body temperature, pressure, and saturated standard convention using the spirometer. Post- bronchodilator spirometry will be performed after 15 to 30 minutes administration of 360 micrograms (4 puffs) of albuterol/salbutamol via metered-dose inhaler.
Percent change from baseline in pre-bronchodilator percent predicted Forced Vital Capacity (FVC) value | Week 1, Week 2, Week 4, Week 8, and Week 12
  FVC will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. FVC is the volume of air that can forcibly be blown out after full inspiration and is measured in liters. Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol.
Percent change from baseline in post-bronchodilator percent predicted Forced Vital Capacity (FVC) value | Week 4 and Week 12
  FVC will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. FVC is the volume of air that can forcibly be blown out after full inspiration and is measured in liters. Post- bronchodilator spirometry will be performed after 15 to 30 minutes administration of 360 micrograms (4 puffs) of albuterol/salbutamol via metered-dose inhaler.
Percent change from baseline in pre-bronchodilator percent predicted Forced Expiratory Flow (FEF) 25-75 value | Week 1, Week 2, week 4, Week 8, and Week 12
  FEF will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. FEF is the speed (or flow) of air coming out of the lung during the middle portion of a forced expiration. It is generally defined by what fraction remains of the forced vital capacity (FVC), usually 25-75 percent (FEF25-75%). Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol.
Percent change from baseline in post-bronchodilator percent predicted Forced Expiratory Flow (FEF) 25-75 value | Week 4 and week 12
  FEF will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. FEF is the speed (or flow) of air coming out of the lung during the middle portion of a forced expiration. It is generally defined by what fraction remains of the forced vital capacity (FVC), usually 25-75 percent (FEF25-75%). Post- bronchodilator spirometry will be performed after 15 to 30 minutes administration of 360 micrograms (4 puffs) of albuterol/salbutamol via metered-dose inhaler.
Percent change from baseline in pre-bronchodilator percent predicted Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) value | Week 1, Week 2, Week 4, Week 8, and Week 12
  FEV1/FVC is the ratio of FEV1 to FVC and will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration and FVC is the volume of air that can forcibly be blown out after full inspiration. Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol.
Percent change from baseline in post-bronchodilator percent predicted Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) value | Week 4 and Week 12
  FEV1/FVC is the ratio of FEV1 to FVC and will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled. FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration and FVC is the volume of air that can forcibly be blown out after full inspiration. Post bronchodilator spirometry will be performed after 15 - to 30 minutes administration of 360 micrograms (4 puffs) of albuterol/salbutamol via metered-dose inhaler.
Change from baseline to Week 12 in Asthma Daily Diary (ADD) data | Week 12
  ADD is an electronic peak flow/diary device to score asthma symptoms twice daily (12 hours interval). Upon awakening, participants are asked to record 3 peak expiratory flow rates (PEFR), number of puffs of albuterol/salbutamol in the past 24 hours and indicate whether they had night time awakenings requiring albuterol/salbutamol. In the evening, participants are asked to record 3 PEFRs and rate asthma symptoms using a 6-point scale (0 = No symptoms and 5 = symptoms so severe that I could not go to work or perform normal daily activities). Higher scores indicate worsening.
Number of participants with worsening of asthma | From baseline (Week 0) to Week 12
  Worsening of asthma is defined as any episode of: 1) decrease in Forced Expiratory Volume in 1 second (FEV1) of greater than or equal to 20 percent compared to baseline FEV1, 2) requiring treatment with systemic corticosteroids, 3) requiring treatment with any other prohibited asthma medication including inhaled corticosteroids, 4) requires emergency room treatment or hospitalization, and 5) life-threatening asthma attack that requires intubation or intensive care unit admission.
Time to worsening of asthma | From baseline (Week 0) to Week 12
Plasma concentrations of JNJ-39758979 | Baseline (Week 0), Week 1, Week 2, Week 4, and Week 12
  Plasma samples will be collected to measure pharmacokintetics of JNJ-39758979.
Serum concentrations of JNJ-39758979 | Baseline (Week 0), Week 1, Week 2, Week 4, and Week 12
  Serum samples will be collected to measure various biomarkers (a substance used as an indicator of a biological state).
Number of participants with adverse events | From screening (Week -6) to Week 17

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (24):
- United States (14):
  - Scottsdale, Arizona
  - Cypress, California
  - Los Angeles, California
  - San Diego, California
  - Normal, Illinois
  - North Dartmouth, Massachusetts
  - Papillion, Nebraska
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Dallas, Texas
  - Waco, Texas
  - Madison, Wisconsin
- Canada (5):
  - Kelowna, British Columbia
  - Niagara Falls, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Québec, Quebec
- India (4):
  - Chennai
  - Mumbai
  - Mysore
  - Pune
- Bucharest, Romania

REFERENCES:
- [Derived] Kollmeier AP, Greenspan A, Xu XL, Silkoff PE, Barnathan ES, Loza MJ, Jiang J, Zhou B, Chen B, Thurmond RL. Phase 2a, randomized, double-blind, placebo-controlled, multicentre, parallel-group study of an H4 R-antagonist (JNJ-39758979) in adults with uncontrolled asthma. Clin Exp Allergy. 2018 Aug;48(8):957-969. doi: 10.1111/cea.13154. Epub 2018 Jun 6. PMID 29682796